CLINICAL TRIAL: NCT04586673
Title: A Phase I Dose Escalation Open Label Trial to Assess Safety and Immunogenicity of Candidate ChAdOx1- and MVA- Vectored Conserved Mosaic HIV-1 Vaccines Given Sequentially to Healthy HIV-1 Negative Adult Volunteers in Oxford, UK
Brief Title: A Study to Assess Safety and Immunogenicity of Conserved Mosaic HIV-1 Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HIV-CORE 0052
Record Dates: First submitted 2020-10-01; First posted 2020-10-14 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2023-08

CONDITIONS: HIV
Keywords: vaccine

STUDY DESIGN:
Intervention Model Description: The first three participants will receive a low dose of ChAdOx1.tHIVconsv1 only. A further ten participants will receive a higher dose of ChAdOx1.tHIVconsv1 and a subsequent vaccination of MVA.tHIVconsv3 and MVA.tHIVconsv4
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChAdOx1.tHIVconsv1 low dose (Experimental): 3 participants will receive one dose of ChAdOx1.tHIVconsv1 at 5 x 10^9 vp
  Interventions: Biological: ChAdOx1.tHIVconsv1 (C1)
- ChADOx1.tHIVconsv1 higher dose (Experimental): 10 participants will receive one dose of ChAdOx1.tHIVconsv1 at 5 x 10^10 vp and one dose each of MVA.tHIVconsv3 at 1 x 10^8 pfu and MVA.tHIVconsv4 at 0.9 x 10^8 pfu.
  Interventions: Biological: ChAdOx1.tHIVconsv1 (C1); Biological: MVA.tHIVconsv3 (M3); Biological: MVA.tHIVconsv4 (M4)

INTERVENTIONS:
Biological: ChAdOx1.tHIVconsv1 (C1) — ChAdOx1.tHIVconsv1 5 x 10^9 vp
  Arms: ChAdOx1.tHIVconsv1 low dose
Biological: ChAdOx1.tHIVconsv1 (C1) — ChAdOx1.tHIVconsv1 5 x 10^10 vp
  Arms: ChADOx1.tHIVconsv1 higher dose
Biological: MVA.tHIVconsv3 (M3) — MVA.tHIVconsv3 1 x 10^8 pfu
  Arms: ChADOx1.tHIVconsv1 higher dose
Biological: MVA.tHIVconsv4 (M4) — MVA.tHIVconsv4 09. x 10^8 pfu
  Arms: ChADOx1.tHIVconsv1 higher dose

SUMMARY:
The object of the study is to assess the safety profile of candidate vaccines ChAdOx1.tHIVconsv1, MVA.tHIVconsv3 and MVA.tHIVcnsv4 administered sequentially in healthy HIV-1/2 negative adult volunteers.

In addition, the study will assess the immune responses generated of the candidate vaccines ChAdOx1.tHIVconsv1, MV.tHIVconsv3 and MVA.tHIVconsv4 administered sequentially in healthy HIV-1/2 negative adult volunteers.

3 healthy, HIV-1 negative adult volunteers will receive one vaccination of low dose ChAdOx1.tHIVconsv1. A further 10 healthy, HIV-1 negative adult volunteers will receive a higher dose of ChAdOx1.tHIVconsv1, followed by one vaccination each of MVA.tHIVconsv3 and MVA.tHIVconsv4 4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-65 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their GP
* Women of child-bearing potential agree to practice continuous effective contraception during the study and test negative for pregnancy on the day(s) of screening and vaccination
* For sexually active men, willingness to use barrier methods for the purposes of contraception from screening until 4 months after the last vaccination
* Agreement to refrain from blood donation during the course of the study
* In the opinion of the Investigators, the volunteer has understood the information provided Written informed consent must be given before any study-related procedures are performed
* Willing to undergo HCV, HBV, syphilis and HIV testing and counselling and receive test results

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant simian adenoviral vaccine prior to enrolment
* Planned receipt of another adenoviral vectored vaccine within 90 days after the vaccination with the ChAdOx1.tHIVconsv1 IMP
* Receipt of any investigational HIV-1/2 vaccine
* Receipt of live attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with the IMP
* Receipt of other vaccine, including influenza vaccine, within the previous 14 days or planned receipt within 14 days after vaccination with the IMP
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV-1/2 infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin)
* History of serious psychiatric condition likely to affect participation in the study
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Reported high-risk behaviour for HIV-1/2 infection. High-risk behaviour for HIV-1/2 infection is defined as follows. Within the previous 12 months the volunteer has:

  * Had unprotected vaginal or anal sex with a person infected with HIV and not taking effective treatment, injecting drug users or casual partners (i.e., no continuing, established relationship)
  * Engaged in sex work for money or drugs
  * Used injection drugs
  * Acquired one of the following sexually transmitted infection: chlamydia, gonorrhea and syphilis.
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Untreated Syphilis: Treponemal IgG/IgM and positive RPR/TPPA AND no documentation of adequate treatment
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cicconi, Principal Investigator — Dr Paola Cicconi
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borthwick N, Fernandez N, Hayes PJ, Wee EG, Akis Yildirim BM, Baines A, Baker M, Byard N, Conway O, Glaze M, Jenkin D, Larkworthy C, Luciw M, Platt A, Poulton I, Thomas M, Quaddy J, Watson M, Crook A, Cicconi P, Hanke T. Safety and immunogenicity of the ChAdOx1-MVA-vectored conserved mosaic HIVconsvX candidate T-cell vaccines in HIV-CORE 005.2, an open-label, dose-escalation, first-in-human, phase 1 trial in adults living without HIV-1 in the UK. Lancet Microbe. 2025 Mar;6(3):100956. doi: 10.1016/j.lanmic.2024.100956. Epub 2024 Nov 26. PMID 39612921

RESULTS

PARTICIPANT FLOW:
Groups:
- ChAdOx1.tHIVconsv1 Low Dose: 3 participants received one dose of ChAdOx1.tHIVconsv1 at 5 x 10^9 vp
  ChAdOx1.tHIVconsv1 (C1): ChAdOx1.tHIVconsv1 5 x 10^9 vp
- ChADOx1.tHIVconsv1 Higher Dose: 10 participants received one dose of ChAdOx1.tHIVconsv1 at 5 x 10^10 vp and one dose each of MVA.tHIVconsv3 at 1 x 10^8 pfu and MVA.tHIVconsv4 at 0.9 x 10^8 pfu.
  ChAdOx1.tHIVconsv1 (C1): ChAdOx1.tHIVconsv1 5 x 10^10 vp
  MVA.tHIVconsv3 (M3): MVA.tHIVconsv3 1 x 10^8 pfu
  MVA.tHIVconsv4 (M4): MVA.tHIVconsv4 09. x 10^8 pfu
Period: Overall Study
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose
Started | 3 | 10
Completed | 3 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: HIV-1/2-negative low risk males and females,18-65 years of age
Groups:
- Total: Total of all reporting groups
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 10 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [32 to 39] | 30 [28 to 37] | 30 [28 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, White British | 3 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Assessement of Safety
Description: • Proportion of volunteers with vaccine related serious adverse events (SAEs) collected up to day 140 after enrollment.
Time Frame: 140 days
Measure: Count of Participants; unit: Participants
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose
Number analyzed (Participants) | 3 | 10
Participants | 0 | 0

2. Primary Outcome: Assement of Safety
Description: Proportion of volunteers with Grade 3 or 4 unsolicited adverse events (AEs) through 28 days post final vaccination
Time Frame: up to 28 days after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose
Number analyzed (Participants) | 3 | 10
Participants | 0 | 6

3. Primary Outcome: Assessment of Safety
Description: Proportion of volunteers with local and systemic reactogenicity events from Day 0 to Day 6 post vaccination
Time Frame: up to day 7
Population: All volunteers were included in the analysis, and all experienced at least one solicited AE after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose
Number analyzed (Participants) | 3 | 10
Participants | 3 | 10

4. Secondary Outcome: Assessment of the Immunogenicity of the ChAdOx1.tHIVconsv1 and MVA.tHIVconsv3 & 4 Vaccines Administered Sequentially.
Description: The proportion of participants that develop T-cell responses to tHIVconsvx measured by IFN-gamma ELISpot assay
Time Frame: Up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose
Number analyzed (Participants) | 3 | 10
Participants | 3 | 10

ADVERSE EVENTS:
Time Frame: Study visits for safety evaluations occurred 1, 7, 14 and 28 days after each vaccination, with additional visits up to days 112 and 140 in Groups 1 and 2, respectively. Safety data included specified, solicited symptoms, collected up to day 7 after each vaccination; unsolicited AEs, collected up to day 28 after each vaccination; and SAEs collected until the end of the study. Blood samples for the evaluation of biochemical and/or haematological parameters were taken at selected study visits.
Description: The severity of clinical and laboratory AEs was assessed according to the scales in the Division of AIDS Table for Grading the Severity of Adult and Paediatric Adverse Events (Corrected Version 2.1, Jul 2017).
Arm/Group | ChAdOx1.tHIVconsv1 Low Dose | ChADOx1.tHIVconsv1 Higher Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChAdOx1.tHIVconsv1 Low Dose (N=3) | ChADOx1.tHIVconsv1 Higher Dose (N=10)
Fatigue (General disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
gastric pain (Gastrointestinal disorders) | 0 | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
warmth at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7) — Local reaction as part of the systematically assessed rectogenicity events
redness at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (10) — Local reaction as part of the systematically assessed rectogenicity events
pain at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (17) — Local reaction as part of the systematically assessed rectogenicity events
itch in injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Local reaction as part of the systematically assessed rectogenicity events
fever (General disorders) | 0 (0) | 2 (3) — Systemic reaction as part of the systematically assessed rectogenicity events
arthralgia (General disorders) | 1 (1) | 8 (10) — Systemic reaction as part of the systematically assessed rectogenicity events
myalgia (General disorders) | 1 (1) | 10 (16) — Systemic reaction as part of the systematically assessed rectogenicity events
feverishness (General disorders) | 2 (2) | 9 (13) — Systemic reaction as part of the systematically assessed rectogenicity events
Headache (General disorders) | 3 (3) | 10 (16) — Systemic reaction as part of the systematically assessed rectogenicity events
Fatigue (General disorders) | 2 (2) | 10 (19) — Systemic reaction as part of the systematically assessed rectogenicity events
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (12) — Systemic reaction as part of the systematically assessed rectogenicity events
Malaise (General disorders) | 2 (2) | 10 (15) — Systemic reaction as part of the systematically assessed rectogenicity events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT04586673/Prot_SAP_000.pdf